CLINICAL TRIAL: NCT00289211
Title: LEVP2005-1/Part A: A Double-blind, Placebo-Controlled, Clinical Study to Investigate the Efficacy and Safety of Purified C1 Esterase Inhibitor (Human) for the Treatment of HAE in Acute Attacks
Brief Title: C1 Esterase Inhibitor (C1INH-nf) for the Treatment of Acute Hereditary Angioedema (HAE) Attacks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEVP2005-1/Part A
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Results first posted 2010-06-02 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary angioedema; HAE; C1 esterase inhibitor (human); C1INH-nf
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C1INH-nf (Experimental): 1,000 Units (U) of C1INH-nf administered intravenously (IV). If there was no response to treatment 60 minutes after the first dose, a second 1,000 U dose could be administered.
  Interventions: Biological: C1 esterase inhibitor [human] (C1INH-nf)
- Placebo (Placebo Comparator): Matching placebo (saline) administered IV. If there was no response to treatment 60 minutes after the first dose, a second placebo (saline) dose could be administered.
  Interventions: Drug: Placebo (saline)

INTERVENTIONS:
Biological: C1 esterase inhibitor [human] (C1INH-nf)
  Arms: C1INH-nf
Drug: Placebo (saline)
  Arms: Placebo

SUMMARY:
The study objective was to determine the safety and efficacy of C1INH-nf for the treatment of acute HAE attacks.

DETAILED DESCRIPTION:
Randomized subjects treated for a qualifying attack were eligible to receive rescue dosing with 1,000 U of C1INH-nf if they did not achieve beginning of substantial relief of the defining symptom within 4 hours after initial treatment with blinded study drug, or if at any time the attack progressed to include airway compromise. A second 1,000 U rescue dose was permitted 60 minutes after the initial rescue dose, if necessary.

The study design also allowed for administration of open-label C1INH-nf for laryngeal angioedema attacks, which were non-randomizable events due to the presence of or potential for airway compromise (immediate 1,000 U dose of C1INH-nf, repeated after 60 minutes, if necessary). In addition, subjects were eligible to receive open-label C1INH-nf (1,000 U single dose) prior to emergency surgical (non-cosmetic) procedures.

A total of 83 subjects were enrolled in the study. Seventy-one (71) subjects experienced qualifying attacks and were randomized to blinded study drug (36 C1INH-nf, 35 placebo); only the 71 randomized subjects were analyzed for efficacy. An additional 12 subjects were never randomized but received open-label C1INH-nf for treatment of laryngeal angioedema and/or prior to emergency surgical procedures. Of the 35 subjects randomized to placebo, 23 also received C1INH-nf (eg, rescue, open-label). In total, 83 subjects received at least 1 dose of study drug and were analyzed for safety; 71 subjects were exposed to C1INH-nf (59 randomized, 12 open-label only) and 12 subjects were exposed only to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Documented HAE
* Normal C1q level

Exclusion Criteria:

* Low C1q level
* B-cell malignancy
* Presence of anti-C1INH autoantibody
* History of allergic reaction to C1INH or other blood products
* Narcotic addiction
* Current participation in any other investigational drug study or within the past 30 days
* Participation in a C1 esterase inhibitor trial, or received blood or a blood product in the past 90 days
* Pregnancy or lactation
* Any clinically significant medical condition, such as renal failure, that in the opinion of the investigator would interfere with the subject's ability to participate in the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-03-14 (Actual); Primary Completion 2007-04-13 (Actual); Study Completion 2007-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (37):
- United States (37):
  - Clinical Research Consultants, Inc, Hoover, Alabama
  - Allergy and Immunology Associates, Scottsdale, Arizona
  - UCLA-David Geffen School of Medicine, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Allergy and Asthma Clinical Research, Inc, Walnut Creek, California
  - Allergy and Asthma Center, Fort Lauderdale, Florida
  - Orlando Regional Healthcare, Orlando, Florida
  - Family Allergy and Asthma Center, Atlanta, Georgia
  - Welborn Clinic Allergy and Immunology, Evansville, Indiana
  - University of Iowa Hospital and Clinic, Iowa City, Iowa
  - The Baton Rouge Clinic, AMC, Baton Rouge, Louisiana
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - Allergy Asthma and Immunology, Falmouth, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Grand Traverse Allergy, Traverse City, Michigan
  - St. Louis University School of Medicine, St Louis, Missouri
  - Nevada Access to Research and Education Society, Las Vegas, Nevada
  - UMDNJ Asthma and Allergy Research Center, Newark, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai School of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - MeritCare Clinical Research, Fargo, North Dakota
  - Bernstein Clinical Research, Cincinnati, Ohio
  - Optimed Research, Columbus, Ohio
  - Allergy Clinic of Tulsa, Tulsa, Oklahoma
  - Allergy Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - Penn State University, Hershey, Pennsylvania
  - Allergy Partners of the Upstate, Greenville, South Carolina
  - AARA Research Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Allergy and Asthma Research Center, San Antonio, Texas
  - Virginia Adult and Pediatric Allergy and Asthma, Richmond, Virginia
  - Marycliff Allergy Specialists, Spokane, Washington
  - Puget Sound Allergy, Asthma and Immunology, Tacoma, Washington
  - Allergy, Asthma and Pulmonary Clinical Research, Madison, Wisconsin

REFERENCES:
- [Derived] Lumry W, Manning ME, Hurewitz DS, Davis-Lorton M, Fitts D, Kalfus IN, Uknis ME. Nanofiltered C1-esterase inhibitor for the acute management and prevention of hereditary angioedema attacks due to C1-inhibitor deficiency in children. J Pediatr. 2013 May;162(5):1017-22.e1-2. doi: 10.1016/j.jpeds.2012.11.030. Epub 2013 Jan 11. PMID 23312695
- [Derived] Grant JA, White MV, Li HH, Fitts D, Kalfus IN, Uknis ME, Lumry WR. Preprocedural administration of nanofiltered C1 esterase inhibitor to prevent hereditary angioedema attacks. Allergy Asthma Proc. 2012 Jul-Aug;33(4):348-53. doi: 10.2500/aap.2012.33.3585. PMID 22856635
- [Derived] Zuraw BL, Busse PJ, White M, Jacobs J, Lumry W, Baker J, Craig T, Grant JA, Hurewitz D, Bielory L, Cartwright WE, Koleilat M, Ryan W, Schaefer O, Manning M, Patel P, Bernstein JA, Friedman RA, Wilkinson R, Tanner D, Kohler G, Gunther G, Levy R, McClellan J, Redhead J, Guss D, Heyman E, Blumenstein BA, Kalfus I, Frank MM. Nanofiltered C1 inhibitor concentrate for treatment of hereditary angioedema. N Engl J Med. 2010 Aug 5;363(6):513-22. doi: 10.1056/NEJMoa0805538. PMID 20818886

RESULTS

PARTICIPANT FLOW:
Groups:
- C1INH-nf: 1,000 Units (U) of C1 esterase inhibitor (C1INH-nf) administered intravenously (IV). If there was no response to treatment 60 minutes after the first dose, a second 1,000 U dose could be administered.
- Open-label C1INH-nf Only: Twelve subjects were never randomized but received open-label C1INH-nf for treatment of laryngeal angioedema and/or prior to emergency surgical procedures. These subjects were analyzed for safety only.
Period: Overall Study
Arm/Group | C1INH-nf | Placebo | Open-label C1INH-nf Only
Started | 36 | 35 | 12
Completed | 36 | 34 | 2
Not Completed | 0 | 1 | 10

BASELINE CHARACTERISTICS:
Groups:
- C1INH-nf: 1,000 U of C1INH-nf administered IV. If there was no response to treatment 60 minutes after the first dose, a second 1,000 U dose could be administered.
- Total: Total of all reporting groups
Arm/Group | C1INH-nf | Placebo | Open-label C1INH-nf Only | Total
Number analyzed (Participants) | 36 | 35 | 12 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (17.68) | 37.0 (13.76) | 36.3 (19.42) | 36.8 (16.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 6 | 61
  Male | 9 | 7 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Time to Beginning of Substantial Relief of the Defining Symptom
Description: Randomized subjects assessed their symptoms every 15 minutes up to 4 hours after the initial dose of blinded study drug or until substantial relief of the defining symptom was achieved. Substantial relief was defined as 3 consecutive assessments of improvement of the defining symptom. Beginning of substantial relief was considered the first of the 3 consecutive assessments.
Time Frame: Within 4 hours after initial treatment
Population: Intent-to-treat (ITT) Population (all randomized subjects). Since less than 50% of subjects in the placebo group achieved the endpoint, median time to event was not estimable (NE). Further, the number of censored events in the C1INH-nf and placebo groups precluded estimation of the 95% confidence interval (CI) upper bound for median time to event.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 36 | 35
hours | 2.0 [1.0 to 4.0] | 4.0 [2.0 to 4.0]
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Subjects who did not experience beginning of substantial relief of the defining symptom within 4 hours after initial treatment were included in the analysis as censored observations. Entries of 4.0 (hours) for median time to event or 95% CI indicate that data were NE (see Population Description). As non-numeric data are not supported by the median and 95% CI fields, entry of the actual results (ie, NE or >4.0) was not possible; Test type: Superiority or Other; p = 0.048, Regression, Cox; Hazard Ratio (HR) = 2.048, 95% CI [1.008 to 4.164]

2. Secondary Outcome: Number of Subjects With Beginning of Substantial Relief of the Defining Symptom
Description: as for outcome 1
Time Frame: Within 4 hours after initial treatment
Population: ITT-Efficacy (ITT-E) Population (N=68; 3 of the 71 randomized [ie, ITT] subjects were excluded from the ITT-E Population, as it was later determined that they did not experience a definitive hereditary angioedema [HAE] attack).
Measure: Number; unit: participants
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 35 | 33
participants | 21 | 14
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.062, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.41, 95% CI [0.87 to 2.29]

3. Secondary Outcome: Time to Complete Resolution of the HAE Attack
Description: Randomized subjects were contacted 72-96 hours (3-4 days) after discharge from the study site to determine when complete resolution of the HAE attack occurred.
Time Frame: 72 hours
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 36 | 35
hours | 12.3 [10.1 to 18.0] | 31.6 [17.8 to 46.0]
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Subjects who had not experienced complete resolution of the HAE attack at the time of the follow-up telephone call, or who were lost to follow-up, were censored at 72 hours; Test type: Superiority or Other; p = 0.001, Regression, Cox; Hazard Ratio (HR) = 2.717, 95% CI [1.471 to 5.020]

4. Secondary Outcome: Antigenic C1 Inhibitor (C1INH) Serum Levels
Description: Change in antigenic C1INH serum levels from pre-infusion to 1-, 2-, 4-, and 12 hours after the initial dose of blinded study drug.
Time Frame: Pre-infusion to 1-, 2-, 4-, and 12 hours post-infusion
Population: ITT-E subjects (N=68) with data available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 35 | 33
mg/dL
  Pre-infusion (N=34, N=33) | 14.7 (22.21) | 13.0 (16.42)
  Change at 1 hour post-infusion (N=35, N=32) | 6.7 (8.86) | -0.9 (9.25)
  Change at 2 hours post-infusion (N=23, N=27) | 11.7 (12.86) | 0.5 (6.73)
  Change at 4 hours post-infusion (N=28, N=23) | 8.6 (8.92) | 0.4 (6.72)
  Change at 12 hours post-infusion (N=19, N=13) | 5.6 (11.21) | -0.8 (4.39)
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Change at 1 hour post-infusion
Statistical Analysis 2: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Change at 2 hours post-infusion
Statistical Analysis 3: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Change at 4 hours post-infusion
Statistical Analysis 4: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.0007, Wilcoxon (Mann-Whitney) — Change at 12 hours post-infusion

5. Secondary Outcome: Functional C1INH Serum Levels
Description: Percent change in functional C1INH serum levels from pre-infusion to 1-, 2-, 4-, and 12 hours after the initial dose of blinded study drug. Functional C1INH serum levels are expressed as a percent of total detectable C1INH (ie, functional C1INH/total detectable C1INH).
Time Frame: Pre-infusion to 1-, 2-, 4-, and 12 hours post-infusion
Population: ITT-E subjects (N=68) with data available.
Measure: Mean (Standard Deviation); unit: percent of functional C1INH
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 35 | 32
percent of functional C1INH
  Pre-infusion (N=34, N=31) | 35.6 (22.62) | 33.7 (29.04)
  Percent change 1 hour post-infusion (N=35, N=32) | 31.5 (23.94) | -6.4 (23.73)
  Percent change 2 hours post-infusion (N=23, N=26) | 45.6 (23.70) | 1.0 (12.43)
  Percent change 4 hours post-infusion (N=28, N=25) | 34.5 (28.22) | 4.3 (26.02)
  Percent change 12 hours post-infusion (N=19, N=14) | 34.8 (17.24) | 5.1 (32.09)
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Percent change 1 hour post-infusion
Statistical Analysis 2: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Percent change 2 hours post-infusion
Statistical Analysis 3: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Percent change 4 hours post-infusion
Statistical Analysis 4: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.0022, Wilcoxon (Mann-Whitney) — Percent change 12 hours post-infusion

6. Secondary Outcome: Complement C4 Serum Levels
Description: Change in complement C4 serum levels from pre-infusion to 1-, 2-, 4-, and 12 hours after the initial dose of blinded study drug.
Time Frame: Pre-infusion to 1-, 2-, 4-, and 12 hours post-infusion
Population: ITT-E subjects (N=68) with data available.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | C1INH-nf | Placebo
Number analyzed (Participants) | 35 | 32
mg/dL
  Pre-infusion (N=35, N=32) | 8.1 (7.79) | 6.7 (5.32)
  Change at 1 hour post-infusion (N=33, N=30) | -0.7 (5.59) | -0.9 (1.96)
  Change at 2 hours post-infusion (N=21, N=26) | -1.7 (8.12) | -1.1 (2.13)
  Change at 4 hours post-infusion (N=26, N=22) | -1.0 (5.62) | -0.5 (1.90)
  Change at 12 hours post-infusion (N=19, N=14) | 2.9 (6.33) | 0.1 (2.07)
Statistical Analysis 1: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.1321, Wilcoxon (Mann-Whitney) — Change at 1 hour post-infusion
Statistical Analysis 2: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.5218, Wilcoxon (Mann-Whitney) — Change at 2 hours post-infusion
Statistical Analysis 3: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.1210, Wilcoxon (Mann-Whitney) — Change at 4 hours post-infusion
Statistical Analysis 4: Comparison: C1INH-nf vs Placebo; Test type: Superiority or Other; p = 0.0017, Wilcoxon (Mann-Whitney) — Change at 12 hours post-infusion

ADVERSE EVENTS:
Time Frame: 3 months. As the study design allowed for all subjects (even those randomized to placebo) to receive C1INH-nf, safety data are presented by actual treatment received (C1INH-nf 71, placebo 12), not randomized treatment group (see Detailed Description).
Description: Presented are all treatment-emergent adverse reactions considered to be related to study drug. There were no serious adverse events reported in this study.
Arm/Group | C1INH-nf | Placebo
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/12
Other Adverse Events (participants affected / at risk) | 2/71 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C1INH-nf (N=71) | Placebo (N=12)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Injection site rash (General disorders) | 1 | 0
Tetany (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement. Most restrictive provision - PI will not publish results until after first of: multicenter publication is published or 24 months from study end. Thereafter, PI may publish his results. PI must provide copy of proposed publication to sponsor for pre-review. If sponsor requests, PI must delete sponsor confidential information before publication and/or delay publication for 90 days so sponsor can file for patents or take other action to protect its patent rights.